CLINICAL TRIAL: NCT00386724
Title: Effectiveness of the Precision Spinal Cord Stimulation System With the Artisan Paddle Electrode in Patients With Back or Lower Extremity Pain
Brief Title: Effectiveness of Precision Spinal Cord Stimulation With Artisan Paddle Electrode
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Data Collected
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCS0406
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Back Pain; Chronic Pain; Pain in Leg, Unspecified
Keywords: Pain; Neurostimulation; Leg Pain; Back Pain
MeSH Terms: conditions — Back Pain; Chronic Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Precision Spinal Cord Stimulation (Experimental): Single arm Precision Spinal Cord Stimulation System with Artisan Surgical Lead
  Interventions: Device: Precision Spinal Cord Stimulation System; Device: Artisan Surgical Lead

INTERVENTIONS:
Device: Precision Spinal Cord Stimulation System — Precision System aids in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with the following: failed back surgery syndrome, intractable back pain, and leg pain.
  Other Names: PRECISION Spinal Cord Stimulator System
Device: Artisan Surgical Lead — Artisan paddle electrode is a 2 x 8 surgical lead approved for use as part of the Precision System.
  Other Names: Artisan surgical lead with PRECISION System.

SUMMARY:
The primary objective of this study is to evaluate the acute and chronic efficacy of spinal cord stimulation using the Precision implantable neurostimulation device with the Artisan paddle electrode in patients with Failed Back Surgery Syndrome (FBSS) and associated primary or secondary back or lower extremity pain. There are significant numbers of patients with FBSS who have moderate to severe drug refractory pain. An optimal outcome will demonstrate that the Precision SCS device has significant effectiveness in reducing this pain resulting in improved quality of life and functional capacity.

DETAILED DESCRIPTION:
The conventional implantation of the spinal cord stimulator calls for dual percutaneous leads placed in parallel at T8-T9 vertebral levels. A common problem after surgery is the migration of leads from the initial implanted site, the consequence of which is inadequate pain relief. Anecdotal reports suggest that the paddle electrode can eliminate some of the problems associated with lead migration by providing a constant distance between the parallel electrodes. Furthermore, it has been reported to provide superior pain relief and paresthesia coverage.

This study aims to evaluate pain and paresthesia coverage by placing a paddle lead. Patients invited to participate in this study will be eligible for SCS therapy and will have already selected therapy with the Advanced Bionics Precision system, independent of possible inclusion in this study.

ELIGIBILITY:
Inclusion Criteria:

* Have FBSS with moderate to severe back or lower extremity pain of at least 3 months duration, be an appropriate candidate for SCS, and have independently elected SCS therapy with the Precision system as next line therapy;
* Be 18 years of age or older;
* Be willing and able to comply with all study related procedures and visits;
* Be capable of reading and understanding patient information materials and giving written informed consent.

Exclusion Criteria:

* Have low back pain as the primary complaint;
* Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints;
* Have participated in any investigational drug or device trial in the last 4 weeks or plan to participate in any other study during the year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Neuromodulation Corporation
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Neurosurgical Specialist, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Precision Spinal Cord Stimulation
Started | 8
3 Months Post-activation | 4
Completed | 3
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Precision Spinal Cord Stimulation
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Baseline Back Pain Severity as Measured at 3 Months Post-activation
Time Frame: 3 months post-activation
Population: The study was terminated and efforts were made to locate data. No study data are available.
Arm/Group | Precision Spinal Cord Stimulation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through completion of study data collection (12 months post-activation or withdrawal)
Arm/Group | Precision Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Precision Spinal Cord Stimulation (N=8)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes